CLINICAL TRIAL: NCT07230782
Title: Percutaneous Ultrasound-Guided Release of the Transverse Carpal Ligament Versus Open Surgery for Carpal Tunnel Syndrome: A Prospective Comparative Study
Brief Title: Ultrasound-Guided Percutaneous Release vs. Open Surgery for Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Principal Investigator, Diego Matías Domínguez Prado, Principal Investigator. Attending phsysician. Orthopaedic Surgeon., Fundacin Biomedica Galicia Sur
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020/580
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Carpal Tunnel Syndrome; Median Neuropathy; Ultrasonography; Surgical Procedures, Operative
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous Ultrasound Guided Release (Experimental)
  Interventions: Procedure: Percutaneous Ultrasound Guided Release of the Transverse Carpal Ligament
- Open surgery (Active Comparator)
  Interventions: Procedure: Open release surgery

INTERVENTIONS:
Procedure: Percutaneous Ultrasound Guided Release of the Transverse Carpal Ligament — A Kemis H3® knife (Newclip, France) with a 12MHz probe were utilized. An 8-10 mm incision was made on the ulnar side of the palmaris longus tendon proximal to the wrist crease. The Kemis H3® knife (Newclip, France) was introduced, with ultrasound visualization ensuring identification and protection of the median nerve and ulnar artery. The flexor retinaculum was sectioned under longitudinal and transverse ultrasound guidance.
  Arms: Percutaneous Ultrasound Guided Release
Procedure: Open release surgery — A short palmar incision (<4 cm) was made along the radial axis of the fourth finger, extending to Kaplan's line. Dissection proceeded to the palmar fascia and flexor retinaculum, which was divided under direct vision and with median nerve protection.
  Arms: Open surgery

SUMMARY:
The goal of this clinical trial is to compare the clinical and functional outcomes of two surgical approaches for the treatment of carpal tunnel syndrome (CTS): ultrasound-guided percutaneous release of the flexor retinaculum and conventional open surgery. The study population includes adults diagnosed with carpal tunnel syndrome who are candidates for surgical treatment.

The main questions this study aims to answer are:

Does ultrasound-guided percutaneous flexor retinaculum release provide superior short-term functional outcomes compared with conventional open surgery?

Does the minimally invasive approach lead to faster symptom relief and postoperative recovery?

Researchers will compare the percutaneous ultrasound-guided technique with the traditional open palmar incision to determine whether the minimally invasive method offers measurable clinical advantages.

Participants will:

Undergo either ultrasound-guided percutaneous release or standard open surgical release, depending on group allocation.

Complete validated clinical and functional assessments at predefined postoperative time points.

Report symptom severity, functional status, and any procedure-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Residence within the hospital's health area
* Clinical and neurophysiological diagnosis of carpal tunnel syndrome
* Underwent surgical treatment between January 2021 and January 2024
* Provided written informed consent for participation and for the publication of anonymized data

Exclusion Criteria:

* Previous surgery for the same pathology in the same hand
* Presence of another associated hand pathology in the same hand
* Patients unable or incapacitated to follow the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Functional outcome measured by the Boston Carpal Tunnel Questionnaire | 3 and 12 months
  The Boston Carpal Tunnel Questionnaire - Symptom Severity Scale and Functional Status Scale, each scored from 1 (no symptoms / no difficulty) to 5 (severe symptoms / inability to perform activities), where higher scores indicate worse clinical symptoms and greater functional impairment.

SECONDARY OUTCOMES:
Pain intensity measured using the Visual Analog Scale | 3 and 12 months
  The Visual Analog Scale for pain (0-10 points), where 0 represents no pain and 10 represents the worst imaginable pain, and higher scores indicate worse pain intensity.
Grip strength measured with a calibrated dynamometer | 3 and 12 months
  Grip strength expressed in kilograms (kg) using a standardized dynamometry protocol. Higher values indicate better hand strength.
Rate of procedure-related adverse events | Intraoperative and up to 12 months postoperative
  Incidence of complications directly attributable to the surgical procedure (e.g., neurovascular injury, pillar pain, infection, incomplete release). Reported as frequency and percentage.
  No scale applicable.
Time to return to normal daily activities | Up to 12 months
  Self-reported number of days required to resume usual daily functions (work, household tasks, leisure). Lower values indicate faster recovery.
Scar-related symptoms and satisfaction | 3 and 12 months
  Assessed using a numeric rating scale from 0 (no symptoms / completely satisfied) to 10 (severe symptoms / completely dissatisfied). Higher scores indicate worse scar-related discomfort or lower satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Alvaro Cunqueiro Hospital, Vigo, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petrover D, Silvera J, De Baere T, Vigan M, Hakime A. Percutaneous Ultrasound-Guided Carpal Tunnel Release: Study Upon Clinical Efficacy and Safety. Cardiovasc Intervent Radiol. 2017 Apr;40(4):568-575. doi: 10.1007/s00270-016-1545-5. Epub 2016 Dec 27. PMID 28028577
- [Background] de la Fuente J, Miguel-Perez MI, Balius R, Guerrero V, Michaud J, Bong D. Minimally invasive ultrasound-guided carpal tunnel release: a cadaver study. J Clin Ultrasound. 2013 Feb;41(2):101-7. doi: 10.1002/jcu.21982. Epub 2012 Sep 11. PMID 22965620
- [Result] Castro-Menendez M, Balvis-Balvis P, Denisiuk M, Vazquez-Cancela O. Assessing the learning curve for percutaneous ultrasound-guided release in carpal tunnel syndrome. J Hand Surg Eur Vol. 2025 Nov;50(10):1365-1370. doi: 10.1177/17531934251338970. Epub 2025 May 8. PMID 40340491

DOCUMENTS (1):
  • Study Protocol (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT07230782/Prot_000.pdf